CLINICAL TRIAL: NCT03341078
Title: Brain Function and Connectivity in Methamphetamine Dependence: The Link to Neuroinflammation and the Effects of Ibudilast
Brief Title: Pilot Study of the Effect of Ibudilast on Neuroinflammation in Methamphetamine Users
Acronym: Ibudilast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Portland VA Medical Center (U.S. Federal Agency); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NURA-001-17F; 16768 (Other: Portland VA Medical Center); 18176 (Other Grant/Funding Number: OHSU); 20053 (Other Grant/Funding Number: OHSU Circle of Giving)
Record Dates: First submitted 2017-10-26; First posted 2017-11-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Methamphetamine-dependence
Keywords: Ibudilast; Methamphetamine; Neuroinflammation
MeSH Terms: conditions — Neuroinflammatory Diseases | interventions — ibudilast

STUDY DESIGN:
Intervention Model Description: Healthy controls will be recruited and have baseline evaluations for neuroinflammation and associated behaviors. Participants with methamphetamine-use disorder will also be recruited and enrolled in a placebo controlled portion of this study. Participants in the placebo controlled portion of this study will be dosed with either the study drug or a placebo twice daily for 6 weeks and will have pre/post evaluations for neuroinflammation and associated behaviors.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Group will be dosed with a placebo oral tablet twice daily for 6 weeks. Participants will have pre/post evaluations for neuroinflammation and associated behaviors
  Interventions: Drug: Placebo Oral Tablet
- Ibudilast (Active Comparator): Ibudilast Group will be dosed with ibudilast twice daily for 6 weeks. The first 2 weeks will be 20 mg twice daily followed by 4 weeks of 50 mg twice daily. Participants will have pre/post evaluations for neuroinflammation and associated behaviors
  Interventions: Drug: Ibudilast
- Controls (No Intervention): Healthy controls will only undergo baseline evaluations and will not be enrolled in the drug portion of the study.

INTERVENTIONS:
Drug: Ibudilast — Ibudilast capsules will be orally ingested twice daily for 6 weeks.
  Arms: Ibudilast
Drug: Placebo Oral Tablet — Placebo capsules will be orally ingested twice daily for 6 weeks.
  Arms: Placebo

SUMMARY:
Addiction to methamphetamine is a serious health problem in the United States. Right now, there are no medications that a doctor can give someone to help them stop using methamphetamine. More research is needed to develop drugs for methamphetamine addiction. Ibudilast (the study drug) is a drug that could help people addicted to methamphetamine.

DETAILED DESCRIPTION:
Addiction to methamphetamine is a serious health problem in the United States. Right now, there are no medications that a doctor can give someone to help them stop using methamphetamine. More research is needed to develop drugs for methamphetamine addiction. Ibudilast (the study drug) is a drug that could help people addicted to methamphetamine.

The investigators are interested to know if the study drug can help some symptoms that methamphetamine can cause, specifically inflammation in the brain. Inflammation has been shown to affect decision-making. The study drug has anti-inflammatory properties, however it is not yet known whether the drug will reduce inflammation in the brain.

ELIGIBILITY:
Inclusion Criteria:

* abstinent from all drugs except marijuana and methamphetamine and have a negative urine drug screen on test days
* Meet diagnosis for recent Methamphetamine-Use Disorder (DSM-V) or does not meet any substance-use disorders

Exclusion Criteria:

* Known sensitivity to ibudilast
* Left handed
* MRI contraindications
* Clinically significant neurological, endocrine, renal, hepatic, or systemic diseases that would compromise safe participation or confound outcomes
* Any psychiatric diagnoses or primary psychotic or mood disorders (past depression diagnoses allowed)
* Any drug use disorder diagnosis besides methamphetamine or tobacco
* Any recreational or prescriptive use of psychotropic medications
* Claustrophobia
* Women who are pregnant or breast-feeding
* Neurodegenerative diseases that present with neuroinflammation
* More than 4 weeks abstinent from methamphetamine
* rs6971 genotype that confers low translocator protein (TSPO) binding affinity to prevent unnecessary radiation exposure
* Liver disease requiring medication or medical treatment and/or aspartate or alanine aminotransferase levels greater than 3 times the upper limit
* Participation in any drug study in the last 3 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Effects of ibudilast on brain function as assessed by magnetic resonance imaging (MRI) | 6 weeks
  Pre and post differences in brain function will be assessed.

SECONDARY OUTCOMES:
Effects of ibudilast on overall cognitive battery score. | 6 weeks
  Pre and post differences in overall cognitive battery score will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Milky Kohno, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2026-01-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03341078/ICF_000.pdf